CLINICAL TRIAL: NCT02756624
Title: A Multi-Center, Double-Masked, Randomized, Vehicle-Controlled, Parallel-Group Study Evaluating the Safety of AC-170 Ophthalmic Solution
Brief Title: A Multi-Center, Vehicle-Controlled, Parallel-Group Study Evaluating the Safety of AC-170 Ophthalmic Solution
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nicox Ophthalmics, Inc. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-100-0010
Record Dates: First submitted 2016-04-20; First posted 2016-04-29 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Cetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AC-170 0.24% (Experimental): 1 drop in each eye 3 times daily for up to 6 weeks
  Interventions: Drug: AC-170 0.24%
- AC-170 Vehicle (Placebo Comparator): 1 drop in each eye 3 times daily for up to 6 weeks
  Interventions: Drug: AC-170 Vehicle

INTERVENTIONS:
Drug: AC-170 0.24%
  Arms: AC-170 0.24%
Drug: AC-170 Vehicle
  Arms: AC-170 Vehicle

SUMMARY:
This is study is evaluating the safety and tolerability of AC-170 Ophthalmic Solution

DETAILED DESCRIPTION:
Central Cornea Endothelial Cell Counts will be done on a subset of approximately 150 subjects to complete 100 subjects as part of the safety measures.

ELIGIBILITY:
Inclusion Criteria:

* at least 2 years of age
* be able to self-administer eye drops or have a parent/legal guardian available for this purpose
* if less than 18 years old have a history or family history of atopic disease (including allergic conjunctivitis)
* have ocular health within normal limits

Exclusion Criteria:

* known contraindications or sensitivities to the study medication or its components
* any ocular condition that, in the opinion of the investigator, could affect the subjects safety trial parameters
* use of disallowed medication during the period indicated prior to the enrollment or during the study
* be pregnant, nursing, or planning a pregnancy

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Protzko, MD, Principal Investigator — Sedeinberg Protzko Eye Associates; Ranjan Malhotra, MD, Principal Investigator — Ophthalmology Associates; Stacey Ackerman, MD, Principal Investigator — Philadelphia Eye Associates; M. Ali Haider, DO, Principal Investigator — Haider Eye Care; Robert Rice, MD, Principal Investigator — R&R Eye Research; Gail Torkildsen, MD, Principal Investigator — Andover Eye Associates
Locations (1):
- Ora Clinical Site Network, Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from six sites in the US.
Pre-assignment Details: There were 516 subjects enrolled, 23 subjects discontinued, and 493 subjects completed the study. Participant flow and baseline characteristics are presented for the 516 subjects that met all inclusion criteria and none of the exclusion criteria and were randomized to receive AC-170 0.24% or AC-170 Vehicle.
Groups:
- AC-170 0.24%: 1 drop in each eye 3 times daily for up to 6 weeks
  AC-170 0.24%
- AC-170 Vehicle: 1 drop in each eye 3 times daily for up to 6 weeks
  AC-170 Vehicle
Period: Overall Study
Arm/Group | AC-170 0.24% | AC-170 Vehicle
Started | 343 | 173
Completed | 327 | 166
Not Completed | 16 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AC-170 0.24% | AC-170 Vehicle | Total
Number analyzed (Participants) | 343 | 173 | 516
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (16.81) | 31.8 (18.3) | 32.2 (17.31)
Age, Customized [Number; unit: participants]
  2-6 years old | 18 | 12 | 31
  2 years old | 6 | 8 | 14
  3 years old | 5 | 2 | 7
  7-12 years old | 29 | 15 | 44
  4-12 years old | 36 | 17 | 53
  13-17 years old | 37 | 17 | 54
  >/= 18 years old | 259 | 129 | 388
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 102 | 299
  Male | 146 | 71 | 217
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 58 | 40 | 98
  Not Hispanic or Latino | 285 | 133 | 418
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 7 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 53 | 32 | 85
  White | 270 | 126 | 396
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 343 | 173 | 516

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of AC 170 0.24% at Visit 1 (Day 1)
Description: Tolerability was assessed upon instillation of study medication, at 1 minute and 2 minutes post study medication instillation. Drop comfort was assessed using a 0-to 10 scale where 0=very comfortable and 10=very uncomfortable.
Time Frame: Upon instillation, 30 Seconds Post-Instillation, 1 minute Post-Instillation
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 Vehicle
Number analyzed (Participants) | 309 | 152
units on a scale
  Upon instillation | 0.87 (1.435) | 0.50 (1.106)
  30 seconds post-instillation | 0.64 (1.181) | 0.42 (0.982)
  1 minute post-instillation | 0.42 (1.001) | 0.31 (0.822)

2. Primary Outcome: Tolerability of AC 170 0.24% at Visit 2 (Day 8)
Description: as for outcome 1
Time Frame: Upon instillation, 30 Seconds Post-Instillation, 1 minute Post-Instillation
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 Vehicle
Number analyzed (Participants) | 299 | 149
units on a scale
  Upon instillation | 0.65 (1.279) | 0.19 (0.665)
  30 seconds post-instillation | 0.38 (0.872) | 0.24 (0.766)
  1 minute post-instillation | 0.26 (0.801) | 0.21 (0.650)

3. Primary Outcome: Tolerability of AC 170 0.24% at Visit 3 (Day 22)
Description: as for outcome 1
Time Frame: Upon instillation, 30 Seconds Post-Instillation, 1 minute Post-Instillation
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 Vehicle
Number analyzed (Participants) | 295 | 148
units on a scale
  Upon instillation | 0.66 (1.321) | 0.43 (1.036)
  30 seconds post-instillation | 0.37 (0.942) | 0.25 (0.725)
  1 minute post-instillation | 0.24 (0.715) | 0.14 (0.446)

4. Primary Outcome: Number of Treatment Related Adverse Events
Description: Adverse events will be measured through study completion
Time Frame: up to 12 weeks
Population: Intent to Treat (ITT)
Measure: Number; unit: adverse events
Arm/Group | AC-170 0.24% | AC-170 Vehicle
Number analyzed (Participants) | 343 | 173
adverse events | 27 | 15

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study. All subjects who received study medication were evaluable for the safety analysis.
Description: Throughout the visits, staff collected all Adverse Events reported, elicited or observed.
Arm/Group | AC-170 0.24% | AC-170 Vehicle
Serious Adverse Events (participants affected / at risk) | 2/343 | 0/173
Other Adverse Events (participants affected / at risk) | 25/343 | 15/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AC-170 0.24% (N=343) | AC-170 Vehicle (N=173)
Substance abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AC-170 0.24% (N=343) | AC-170 Vehicle (N=173)
Visual acuity reduced (Eye disorders) | 4 (5) | 4 (4)
Conjunctival hyperemia (Eye disorders) | 4 (4) | 3 (3)
Punctate keratitis (Eye disorders) | 3 (3) | 3 (3)
Instillation site pain (General disorders) | 6 (7) | 1 (1)
Instillation site erythema (General disorders) | 0 (0) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes